CLINICAL TRIAL: NCT00187148
Title: Evaluation of the Tolerability and Safety of a Recombinant HIV-1 Multi-Envelope DNA Plasmid Vaccine (EnvDNA) in Healthy Adults
Brief Title: Evaluate Tolerability of a Recombinant DNA HIV-1 Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EnvDNA; IND11130
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2011-06

CONDITIONS: Human Immunodeficiency Virus; HIV Infections
Keywords: Vaccine; Prevention; HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Biological: EnvDNA

INTERVENTIONS:
Biological: EnvDNA — administered as 100 mcg of DNA in 1.5mL PBS every 28 days for 3 injections

SUMMARY:
This protocol will evaluate the safety and tolerability of the vaccine EnvDNA in healthy adults. DNA-based vaccines are being studied for the prevention of human immunodeficiency virus (HIV), malaria and hepatitis. DNA vaccines have been well tolerated in human studies to date. The vaccine that will be tested in this study was made from the information that the virus uses to make a small part of the HIV. This small part is called the envelope or coating around the virus. We hope the body will make an immune response against the HIV envelope coat. Our potential HIV DNA envelope vaccine is called EnvDNA.

DETAILED DESCRIPTION:
This is a research (investigational) study to find out about the safety of a new potential vaccine for HIV. This potential vaccine may eventually become a part of a sequence of three experimental vaccines that will be studied to see if they can help to protect people from HIV. HIV infection is the cause of AIDS (Acquired Immune Deficiency Syndrome). AIDS is one of the most serious viral infections we know. This study is being done to help us find an HIV vaccine that works.

The vaccine that will be tested in this study was made from the information that the virus uses to make a small part of the HIV. This small part is called the envelope or coating around the virus. Because only the information for this one part of the virus is used in the vaccine, the vaccine cannot cause HIV infection. We make the vaccine in a test tube. The vaccine is made up of DNA. DNA is like an instruction manual that cells use to make basic building blocks called proteins. This DNA has the information that cells will use to make the envelope coat of HIV. Once the DNA is injected intramuscularly, it should tell cells to make the envelope protein. We hope the body will make an immune response against the HIV envelope coat. Our potential HIV DNA envelope vaccine is called EnvDNA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults; age greater than 18 years, less than or equal to 40 years
* HIV-1 negative as documented by negative ELISA and negative Western blot analysis within 30 days prior to immunization
* Normal history and physical exam
* Normal complete blood count and differential obtained within 60 days prior to immunization, and defined as:

  * hemoglobin greater than or equal to 12.0 gm/dl for females and greater than or equal to 14.0 gm/dl for males
  * white blood cell count greater than or equal to 3500 cells/mm3
  * platelet count between 150,000 and 550,000 cells/mm3
  * CD4+ T cell count greater than or equal to 400 cells/mm3 (if a single CD4+ T cell count <400 cells/mm3 is obtained, a repeat count will be performed and immunization will proceed if the repeat count is greater than or equal to 400 cells/mm3)
* Anti-nuclear antibody titer <1:80 (by IFA) and negative anti-DNA antibody within 60 days prior to immunization
* Negative for Hepatitis B surface antigen and Hepatitis C
* AST and ALT within normal institutional limits obtained within 60 days prior to immunization
* Serum creatinine, Na+, K+ and Cl- within normal institutional limits, obtained within 60 days prior to immunization
* Serum creatine phosphokinase (CPK) within normal institutional limits obtained within 60 days prior to immunization
* Not planning to become pregnant during study vaccinations and for three months after last vaccination
* Availability for at least one year of follow-up

Exclusion Criteria:

* History of immunosuppressive illness, chronic illness (e.g. asthma, diabetes, hypertension, bleeding diathesis, etc), or
* Receiving therapy or prophylaxis for tuberculosis
* Medical or psychiatric condition or occupational responsibilities which preclude subject compliance with the protocol. Specifically excluded are persons with a history of suicide attempts, recent suicidal ideation or who have past or present psychosis
* Live attenuated vaccines within 60 days of study enrollment (Note: subunit or killed vaccines [e.g. influenza or pneumococcal] are not exclusionary, but should be given at least 2 weeks before or after HIV immunization)
* Use of experimental agents within 30 days prior to study enrollment
* Receipt of blood products or immunoglobulin in the past 6 months
* Subjects with known allergy to the antibiotic kanamycin
* Pregnancy at the time of vaccination (urine pregnancy test)
* Nursing mother at the time of vaccination
* Any member of the Investigator's laboratory program
* Participation in previous HIV vaccine trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2005-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the tolerability and safety of the EnvDNA vaccine | 1 year

SECONDARY OUTCOMES:
To characterize the kinetics, duration and magnitude of any HIV-envelope specific immune response elicited by EnvDNA | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pat Flynn, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org